CLINICAL TRIAL: NCT03225976
Title: Effect of Light-Emitting Diode on the Strenght and Resistence Capacities of Cycling Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rinaldo Roberto de Jesus Guirro, Professor Doctoral, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: U1111-1143-7629
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Athletes
Keywords: Phototherapy; Athletic Performance; Muscle Strength; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: Athletes will be randomized allocated the following groups:
  * Infrared LED group (G-I; n = 12)
  * Red LED group (G-V; n = 12)
  * Infrared plus Red LED group (G-IV; n = 12)
  * Sham Group (G-S; n = 12)
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Infrared LED group (G-I) (Experimental): The Light-Emitting Diode Device with wavelength of 904nm will be applied throughout the quadriceps femoralis extension bilaterally.
  Interventions: Device: Light-Emitting Diode Device
- Red LED group (G-V) (Experimental): The Light-Emitting Diode Device with a wavelength of 620nm will be applied throughout the quadriceps femoralis extension bilaterally.
  Interventions: Device: Light-Emitting Diode Device
- Sham Group (G-S) (Sham Comparator): The Sham Light-Emitting Diode Device will be positioned throughout the quadriceps femoral muscle extension, however, there will be no light emission.
  Interventions: Device: Sham Light-Emitting Diode Device
- Infrared plus Red LED group (G-IV) (Experimental): The Light-Emitting Diode Device with a wavelength of 620nm plus 904nm will be applied throughout the quadriceps femoralis extension bilaterally.
  Interventions: Device: Light-Emitting Diode Device

INTERVENTIONS:
Device: Light-Emitting Diode Device — The therapy will be applied on the second, third and fourth day of collection using a 25x40 cm2 LED blanket, with an equidistant distribution, with total energy per area of 180 J bilaterally on the quadriceps femoris muscle.
  All LEDs will be calibrated prior to the start of applications in the Laboratory of Photobiophysics of the Faculty of Sciences and Letters of Ribeirão Preto, University of São Paulo, in which the wavelengths will be checked, the angle of radiation, power and power density.
  Arms: Infrared LED group (G-I); Infrared plus Red LED group (G-IV); Red LED group (G-V)
Device: Sham Light-Emitting Diode Device — The Sham Light-Emitting Diode Device will be applied on the second, third and fourth day of collection using a 25x40 cm2 LED blanket, with an equidistant distribution, with total energy per area of 0 J bilaterally on the quadriceps femoris muscle. At the time of application the device will not be activated
  Arms: Sham Group (G-S)

SUMMARY:
Phototherapy is a therapeutic resource of increasing use in the last decade. The photobiomodulatory effects are commonly produced by means of low intensity lasers or LED emitting diodes, and can be used at different wavelengths. These light sources are divergent as to coherence, but produce equivalent tissue effects. The application of laser or LED light is able to induce biochemical changes in tissues, allowing for inhibitory or stimulating effects. These responses are associated to a cascade of cellular reactions, which favor the absorption of enzymes by cytochrome c oxidase, generating physiological responses that lead to decreased production of reactive oxygen species and increased synthesis of adenosine triphosphate (ATP). The application of this therapeutic resource brings ergogenic and protective benefits in muscular performance. The use of LED as a light source is promising because of its low cost, but there are no enough studies that support this use in athletes, with a focus on performance improvement. In addition to the deficiency of the sample, there is also no consensus regarding the use of different wavelengths for LED in the literature, thus opening gaps for the best protocol for the application of this technique. Therefore, a study that evaluates the use of LED in athletes, with different wavelengths, to improve performance is necessary. Hypothesis: It is hypothesized that the LED application is capable of improving athletes performance in terms of increased fatigue resistance, increased strength and power, increased muscle recruitment, and optimized oxygen demand. It is also expected that the results generated in this study can contribute to and increase the resources used by physiotherapists within the clinical-sports field, contributing to the post-training recovery, as well as the more effective physical performance in competitive activities.

DETAILED DESCRIPTION:
Background: Phototherapy is a therapeutic resource of increasing use in the last decade. The photobiomodulatory effects are produced by sources of low-level lasers or light- emitting diode (LEDT), and their tissue effects are equivalent. The application of this therapeutic resource brings ergogenic and protective benefits in muscular performance. The use of LED as a light source is promising because of its low cost, but there are no enough studies that support this use in athletes, with a focus on performance improvement. In addition to the deficiency of the sample, there is also no consensus regarding the use of different wavelengths for LED in the literature, thus opening gaps for the best protocol for the application of this technique. Therefore, a study that evaluates the use of LED in athletes, with different wavelengths, to improve performance is necessary. Objective: To analyze the acute effects of the application of LED phototherapy on the strength and fatigue strength abilities of cycling athletes. Method: The study sample will be composed of 48 male cyclist athletes randomly allocated into three groups: Infrared LED Group (G-I), Red LED Group (G-V), Infrared plus Red Group (G-IV) and Sham Group (G-S). The athletes will be submitted to a battery of tests, for performance evaluation which consist of anaerobic and aerobic power and threshold, bioimpedance, infrared thermography, creatine kinase (CK) and blood lactate analysis, measurement of local muscle blood flow, Gas analysis, besides the isokinetic, electromyographic and biomechanical evaluations. After 24 hours of the tests, the LEDT (180 J) will be applied three times in three differents days to the quadriceps femoris muscle bilaterally. The same tests will be performed 24 hours after the application of LEDT. In the 1st and 4th week, post intervention, only the isokinetic and electromyographic evaluations will be performed. For analysis of the data, normality test will be used to verify the distribution and adequate statistical tests for the appropriate intra and intergroup comparisons, being considered two factors in the comparisons, time and group. A significance level of 5% will be adopte

ELIGIBILITY:
Inclusion Criteria:

* Cycling practitioners
* Age between 18 and 45 years;
* Male
* VO2MÁX > 40 ml.kg-1.min-1;
* Absence of musculoskeletal injury in the last six months

Exclusion Criteria:

* Carriers of Cardiorespiratory Diseases;
* Users of anti-inflammatory and analgesic drugs
* Users of Alcohol and illicit drugs

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-12-25 (Actual); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
Strenght Capacities | Twenty minutes
  N/m

SECONDARY OUTCOMES:
Resistence Capacities | Twenty Minutes
  Minutes
Muscle recruitment | Twenty Minutes
  Hertz
Gas analysis | Twenty Minutes
  ml.kg-1.min-1
Lactate analysis | Twenty Minutes
  mmol/L
Creatine Kinase Analysis | Five Minutes
  IU/L
Thermography | Fifteen Minutes
  Celsius Degree
Local blood flow | Twenty Minutes
  mL/s
Power | Twenty Minutes
  Watts

CONTACTS AND LOCATIONS:
Overall Officials: Rinaldo RJ Roberto de Jesus Guirro, Dr, Study Director — University of Sao Paulo
Locations (1):
- University of São Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ferraresi C, Huang YY, Hamblin MR. Photobiomodulation in human muscle tissue: an advantage in sports performance? J Biophotonics. 2016 Dec;9(11-12):1273-1299. doi: 10.1002/jbio.201600176. Epub 2016 Nov 22. PMID 27874264
- [Derived] de Carvalho G, Gobbi A, Gobbi RB, Alfredo DMN, do Carmo Furquim TH, Barbosa RI, Papoti M, de Jesus Guirro RR. Photobiomodulation by light emitting diode applied sequentially does not alter performance in cycling athletes. Lasers Med Sci. 2020 Oct;35(8):1769-1779. doi: 10.1007/s10103-020-02973-9. Epub 2020 Feb 20. PMID 32078062
- See also: Page intended to research scientific articles published in journals — https://www.ncbi.nlm.nih.gov/pubmed/